CLINICAL TRIAL: NCT02013011
Title: Effects of Recruitment Maneuver in Patients Undergoing Robotic Assisted Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-1306/206-004
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2014-07

CONDITIONS: Effects of Recruitment Maneuver During Intraoperative and Postoperative Period

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- recruitment maneuver and PEEP (Active Comparator): apply recruitment maneuver and positive end expiratory pressure (PEEP) 5 centimeter of water (cmH2O) after induction of anesthesia
  Interventions: Procedure: recruitment maneuver(RM) and positive end expiratory pressure(PEEP) or PEEP only
- PEEP (Active Comparator): apply positive end expiratory pressure (PEEP) 5 cmH2O after induction of anesthesia
  Interventions: Procedure: recruitment maneuver(RM) and positive end expiratory pressure(PEEP) or PEEP only

INTERVENTIONS:
Procedure: recruitment maneuver(RM) and positive end expiratory pressure(PEEP) or PEEP only — application of recruitment maneuver(RM) and positive end expiratory pressure(PEEP) in RM and PEEP group and application of only PEEP in PEEP group

SUMMARY:
This study is to evaluate effects of recruitment maneuver in patients undergoing robotic assisted radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* 60~80 yr
* American Society of Anesthesiologists physical status 1 or 2
* scheduled for elective robotic assisted radical prostatectomy

Exclusion Criteria:

* heavy smoker
* severe respiratory or cardiac disease
* hepatic or renal function impairment
* neurologic disease
* BMI > 31kg/m2

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
rate of perioperative complication | perioperative period
  check the rate of perioperative complication( desaturation during operation and postoperative atelectasis in each groups

SECONDARY OUTCOMES:
respiratory index | intraoperative respiratory index
  static & dynamic compliance, results of arterial blood gas analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Ah-young Oh, Seongnam-si, Gyeonggi-do, South Korea